CLINICAL TRIAL: NCT02162940
Title: Effect of Statin Use on Low Back Pain Steroid Injections.
Brief Title: Statin and Epidural Steroid Injection
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, MD, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: SARI-06
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain After Epidural Steroid Injection; Quality of Life After Epidural Steroid Injection
Keywords: low back pain; epidural steroid injection; statin; quality of life
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients taking statins: Visual anlogue score vas used to evaluate pain. The SF 36 test was used to evaluate quality of life.
  Interventions: Other: Visual analogue score; Other: The SF 36 test
- patients not taking statins: Visual anlogue score vas used to evaluate pain.The SF 36 test was used to evaluate quality of life.
  Interventions: Other: Visual analogue score; Other: The SF 36 test

INTERVENTIONS:
Other: Visual analogue score — Visual analogue score vas used to evaluate pain.
  Other Names: VAS score
Other: The SF 36 test — The SF 36 test (SHORT FORM 36) was used to evaluate quality of life.
  Other Names: SHORT FORM 36

SUMMARY:
The impact of statin use on response to epidural steroid injections remains unknown and may well increase the effect considering the substantial anti-inflammatory properties. We thus tested the primary hypothesis that patients taking statins before and after the procedure will have lower VAS scores compared to patients not on statins. Secondarily we tested the hypothesis that statin users will have improved quality of life evaluated with Short Form 36 (SF 36).

DETAILED DESCRIPTION:
Low back pain is one of the most common complaints for physician office visits and is the most common disorder requiring interventional pain treatment in USA. Fluoroscopy-assisted transforaminal anterior epidural steroid injections (TAESI) are more commonly preferred for treatment of low back pain. Most of the time epidural steroid injections are supplemented with different analgesic combinations due to insufficient analgesia. Recent reports have revealed immunomodulatory and anti-inflammatory activities for statins in vivo and in vitro. Statins have very recently been shown to alleviate neuropathic pain in the rat model. However, the impact of statin use on response to epidural steroid injections remains unknown and may well increase the effect considering the substantial anti-inflammatory properties. We thus tested the primary hypothesis that patients taking statins before and after the procedure will have lower VAS scores compared to patients not on statins. Secondarily we tested the hypothesis that statin users will have improved quality of life evaluated with Short Form 36 (SF 36).

ELIGIBILITY:
Inclusion Criteria:

* indication for TAESI given by blinded pain physician

Exclusion Criteria:

* known allergy to steroids
* indication for surgery
* unstable opioid use
* drug or alcohol abuse within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients coming to the Algology Department with complaints of low back pain and scheduled to receive Transforaminal epidural steroid injection. Statin users (Group 1) and non-statin users (Group 2) will be record.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Low back pain after transforaminal epidural steroid injection assessed by VAS scale. | 6 months

SECONDARY OUTCOMES:
Quality of life was evaluated with SF 12 test. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Osman Nuri Aydın, Prof, Principal Investigator — Adnan Menderes University Medical Faculty Algology Department; Banu Taşdemir, Asist Dr, Principal Investigator — Adnan Menderes University Medical Faculty Anesthesiology and Reanimation Department; Fabrizio Galimberti, Medical Student, Principal Investigator — Cleveland ClinicLernerCollege of Medicine, Cleveland, Ohio; Alparslan Turan, Associate Prof, Principal Investigator — Department of Outcomes Research, Cleveland Clinic; Sinem Sari, Assist Prof, Study Chair — Adnan Menderes University Medical Faculty Anesthesiology and Reanimation Department
Locations (1):
- Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin, Turkey (Türkiye)

REFERENCES:
- [Result] Gillon JT, Smith SE, Lowden MR. Atorvastatin as novel treatment for neuropathic pain: a case report. Clin J Pain. 2013 Dec;29(12):e46-8. doi: 10.1097/AJP.0b013e3182a03c2e. PMID 23887344